CLINICAL TRIAL: NCT06916520
Title: Prasugrel Monotherapy Reduced Dose in Acute and Chronic Coronary Syndrome Patients After Percutaneous Coronary Intervention
Brief Title: Prasugrel Monotherapy Reduced Dose in Acute and Chronic Coronary Syndrome Patients After Percutaneous Coronary Intervention (PROMOTE)
Acronym: PROMOTE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: J.P.S Henriques (Other)
Responsible Party: Sponsor-Investigator, J.P.S Henriques, Professor Doctor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMOTE; 2024-520351-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Coronary Arterial Disease (CAD); Percutaneous Coronary Intervention (PCI)
MeSH Terms: interventions — Prasugrel Hydrochloride; 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Prasugrel low-dose monotherapy
  Interventions: Drug: Prasugrel 5 mg
- Control Arm (Active Comparator): Dual antiplatelet therapy
  Interventions: Drug: Dual Antiplatelet (DAPT) Therapy

INTERVENTIONS:
Drug: Prasugrel 5 mg — Prasugrel 5 mg once daily (monotherapy)
  Arms: Intervention Arm
Drug: Dual Antiplatelet (DAPT) Therapy — Dual antiplatelet therapy according to guidelines
  Arms: Control Arm

SUMMARY:
Rationale: Dual antiplatelet therapy, consisting of aspirin and a P2Y12-inhibitor, reduces the risk of stent-related and non-stent-related ischemic events after percutaneous coronary intervention (PCI). However, this therapy is also associated with a higher risk of bleeding. Given the advances in stent technology and pharmacology, it may be possible to treat patients undergoing PCI with low dose prasugrel as single antiplatelet therapy, regardless of medical history, age or body weight.

Objective: Assess the feasibility and safety of a single antiplatelet strategy with a reduced dose of prasugrel 5 mg after PCI in acute and chronic coronary syndrome patients (ACS and CCS).

Study design: Open-label, single-centre, randomized controlled trial pilot.

Study population: Patients undergoing successful PCI due to acute or chronic coronary syndrome.

Intervention: A once-daily reduced dose of 5 mg prasugrel for 6 months in CCS patients and for 12 months in ACS patients, preceded by a loading dose of 60 mg prasugrel after PCI, administered without concomitant use of aspirin.

Main study parameters/endpoints: The primary endpoint is Net Adverse Clinical Events (NACE), a composite of all-cause death, myocardial infarction, definite stent thrombosis, ischemic stroke, clinically relevant non-major bleeding or major bleeding defined as Bleeding Academic Research Consortium type 2, 3 or 5.

ELIGIBILITY:
Inclusion Criteria:

* Acute Coronary Syndrome
* Chronic Coronary Syndrome
* Successful PCI

Exclusion Criteria:

* Known allergy or contraindication for prasugrel, including Active pathological bleeding Severe liver disease (defined as Child Pugh class C)
* Current indication for oral anticoagulant therapy (OAC)
* Indication for ongoing DAPT (e.g. PCI ≤ 6 months for CCS or ACS ≤ 12 months)
* Pregnancy or breast-feeding women
* Participation in another trial with an investigational drug or device
* Recent or ongoing strong CYP3A4 inhibitor or inducer therapy (e.g. clarithromycin, ketoconazole, carbamazepine or rifampicin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
NACE (Net Adverse Clinical Events) | 12 months
  The primary endpoint is NACE, a composite of all-cause mortality, myocardial infarction, definite stent thrombosis, ischemic stroke, major bleeding or clinically relevant non-major bleeding defined as BARC type 2, 3 or 5

IPD SHARING:
Plan to Share IPD: Undecided